CLINICAL TRIAL: NCT01567982
Title: Phase 1 Study of Effects of tDCS on Tobacco Withdrawal Symptoms
Brief Title: Effects of Transcranial Direct Current Stimulation on Tobacco Withdrawal Symptoms
Acronym: tDCSsmokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jiansong Xu, Assistant Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1008007212; K01DA027750 (NIH)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Nicotine Withdrawal; Tobacco Abstinence
Keywords: tDCS; brain stimulation; addiction; substance dependence; craving; cognition
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- smokers and nonsmokers (Experimental): both smokers and nonsmokers will receive same tDCS
  Interventions: Device: tDCS, prefrontal cortex and parietal cortex

INTERVENTIONS:
Device: tDCS, prefrontal cortex and parietal cortex — tDCS is a non invasive brain stimulation methods. We will use two anodes to stimulate prefrontal and/or parietal cortex using 2mA current for 20 minutes.
  Other Names: transcranial direct current stimulation

SUMMARY:
We hypothesize that transcranial direct current stimulation will reduce tobacco withdrawal symptoms of tobacco dependent smokers abstinent from smoking for more than 10 hours.

DETAILED DESCRIPTION:
We will recruit 35 non-smokers and 30 adult smokers who smoke > 15 cigarettes/day for more than two years and are 18-55 years old. We expect about half of them will be females. All participants will be screened for drugs of abuse and female participants will receive a pregnancy test. Each smoker will participate in four tDCS sessions, one for sham and three for real tDCS, each for one set of electrode montage. The first set is dorsal lateral prefrontal cortex (i.e., F3 and F4 of 10/20 EEG system) and neck. The second set is middle line prefrontal cortex (Fz), superior parietal cortex (Pz), and bilateral inferior temporal cortex (T3 and T4). The third set is left dorsal lateral prefrontal cortex (F3) and superior parietal cortex (P1), and right inferior temporal cortex (T4). The sequence of real and sham tDCS will be counterbalanced among participants. Each session will last for 20 minutes and there will be a minimum 48 hours between the two sessions. Participants will be required to be abstinent from cigarette smoking overnight for a minimum of 10 hours and arrive at our lab around 8:30 AM for each tDCS session. After arrival, each participant will provide a breath sample for detection of any alcohol in their system, an assay of CO and for verification of abstinence from cigarette smoking. We will place a nicotine patch (Nicoderm with 21 mg nicotine) on the back of participants. We will also ask each participant to chew a nicotine gum (Nicorette gum with 4 mg nicotine) for 30 minutes. The participants will perform a battery of computerized tasks including the N-Back working memory task, and an attention task involving watching a computer screen and pressing buttons to indicate more odd or even numbers displayed on the screen. In addition participants will complete the following questionnaires related to mood, nicotine withdrawal, mental state, possible side effects, and cigarette craving: Profile of Mood States (McNair et al 1971), Shiffman-Jarvik Withdrawal Scales (Shiffman & Jarvik 1976), and Urge To Smoke (Jarvik et al 2000), tDCS side effects questionnaire, Wisconsin Smoking Withdrawal Scale (Welsch 1999), Perceived Stress Scale (Cohen 1983), Spielberger State/Trait Anxiety Questionnaire (Spielberger 1970).

Each participant will repeat above battery of cognitive tasks and questionnaires after tDCS. Then they will be instructed to smoke one cigarette after this second battery of tasks/questionnaires, and repeat the second battery of questionnaires after cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Age between 18 and 55 yrs
* Smokers must smoke at least 15 cigarettes per day for the past two years (as indicated by self-report)
* Must give a breath CO sample of at least 15 ppm to verify current tobacco consumption during screen
* Must give a breath CO sample of 7 or less ppm to verify tobacco abstinence during the abstinence session
* Cocaine and alcohol patients should meet DSM-IV criteria, and is confirmed after clinical interview with a structured interview with the SCI-PG and SCID-P.
* Right-handed, as indicated by the Edinburgh Handedness Questionnaire
* Smokers should have no illicit drug use, as indicated by negative results on urine drug screens of cocaine, methamphetamine, opiates, or benzodiazepines at all sessions
* Smokers should consume less than or equal to 10 standard drinks of alcohol per week (one standard drink consists of one 12 oz. beer, 6 oz. of wine, or one shot (1.5 oz.) of hard liquor (80 proof) (as indicated by self-report)
* Absence of any past or current DSM-IV Axis I diagnoses (as verified by the SCID)
* English as a first language (subjects may be bilingual), and able to read and speak English fluently (as indicated by self-report)

Exclusion Criteria:

* Any medically significant acute or chronic medical condition as indicated by self-report (significance is determined by the P.I.)
* English as a second language (as indicated by self-report)
* Left-handed or ambidextrous as indicated on the Edinburgh Handedness Questionnaire
* Marijuana use of greater than one joint once per week. The subject's urine must screen negative at each session, so the subject is instructed to refrain from using marijuana for the 72 hours prior to each session.
* Pregnant, as indicated by a positive result on the urine pregnancy test given at each session
* Below normal intelligence (Shipley estimated IQ of 85 or less) as indicated by a combined score of <45 on the Shipley Institute of Living Scale
* Evidence of head injury involving loss of consciousness for 5 minutes or more and/or requiring hospitalization (as indicated by self-report)
* Depression, as assessed by the SCID or a score of >18 on the BDI (see appendix)
* Probable childhood ADHD as indicated by a score of >46 on the Wender Utah Rating Scale and/or by self-report
* Self-report of learning disability or dyslexia
* Current or past use of psychotropic drugs (i.e., any antidepressants, antipsychotics, psychostimulants (i.e. Ritalin), benzodiazepines (i.e., Valium, Xanax), or use of any other drugs known to affect cognitive functioning (as indicated by self-report).
* HIV positive (as indicated by self-report)
* Positive TB test (as indicated by self-report)
* For subjects participating in the smoking portion, consumption of more than 10 standard drinks of alcohol per week (see inclusion criteria for description of standard drink)
* Presence of any past or current DSM-IV Axis I Diagnoses, as verified by the SCID
* Abnormal uncorrected vision or hearing which would affect performance on cognitive tests (as indicated by self-report)
* Smokers group:
* Has not smoked 15 or more cigarettes per day for a minimum of the past 2 years
* A CO breath sample of <15 ppm during any session (except the abstinence session)
* Presence of a pacemaker, catheter or device implant that might be interfered with by the current applied during tDCS.

  b) Eligibility to participate in the study will be determined by trained research personnel who will screen potential participants over the phone.

  c) Minors are excluded because the study involves cigarette smoking. Participants over 55 are excluded due to their increased probability of smoking-related and age-related health problems. Pregnant women or those of childbearing potential who are not using birth control will be excluded because the studies involve cigarette smoking and therefore pose a risk to a fetus.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Urge to Smoke scale | 20 minutes
  This is a 10-item self-report questionnaire. It measures the level of urge to smoke cigarette
Negative affect | 10 min
  Use self-report questionnaire Profile of Mood States to assess negative affect

SECONDARY OUTCOMES:
Reaction time on an attention task | 20 minutes
  Participants will perform a computerized visual attention task. Performance measures including reaction time and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansong Xu, Ph.D., Principal Investigator — Yale University
Locations (1):
- 1 Church Street, Room 729, New Haven, Connecticut, United States